CLINICAL TRIAL: NCT03498729
Title: The Role of Autoimmune Mechanisms in the Pathogenesis of Atrial Fibrillation
Brief Title: Autoimmunity in the Pathogenesis of AF
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Rowlens M. Melduni, Consultant, Mayo Clinic
Other Study IDs: 16-005678; 1K01HL135288-01 (NIH)
Record Dates: First submitted 2017-11-19; First posted 2018-04-17 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Atrial Fibrillation
Keywords: Autoimmune Diseases
MeSH Terms: conditions — Atrial Fibrillation; Autoimmune Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Persistent AF
  Interventions: Other: Peripheral Blood Sample
- Paroxysmal AF
  Interventions: Other: Peripheral Blood Sample
- Psoriasis
  Interventions: Other: Peripheral Blood Sample
- Healthy Controls
  Interventions: Other: Peripheral Blood Sample

INTERVENTIONS:
Other: Peripheral Blood Sample — 30mL peripheral whole blood sample

SUMMARY:
This research study is being done to find out whether autoimmune mechanisms are associated with the development of atrial fibrillation.

DETAILED DESCRIPTION:
The study sets out to identify an explanation for the pathogenesis of AF, potentially forming the basis for designing novel targeted therapies to prevent or reverse this prevalent human disease. The overall objectives are to determine whether autoimmune diseases are associated with AF development and to identify specific diagnostic and prognostic biomarkers that will improve the ability to accurately predict risk of AF development. The study will prospectively enroll patients with and without AF and determine their serum cytokine levels and assess the functional responses of T cells on the basis of cytokine production after in vitro T-cell specific stimulation, using Luminex bead-based multiplex technology.

ELIGIBILITY:
Inclusion Criteria:

* Cases: AF (Persistent, paroxysmal AF)
* Controls 1: (No prior history of AF or inflammatory or autoimmune diseases)
* Controls 2: (biopsy proven Psoriasis)

Exclusion Criteria:

* Clinically apparent acute infections over the past 4 weeks
* Chronic infections
* Recent malignancies
* Recent Radiation or chemotherapy
* Chronic kidney disease (≥ stage 2)
* Organ transplantation
* History of chronic liver disease
* Major surgery or invasive procedure in the past 6 months
* Internal prosthesis
* Receiving immunosuppressive therapy
* Known rheumatologic diseases (except for the participants with psoriasis)
* Females who are known to be pregnant

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients 18 years and older.
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2021-12-09 (Actual); Study Completion 2021-12-09 (Actual)

PRIMARY OUTCOMES:
Cytokines Levels | through study completion, approximately 3 years.
  Cytokine Profiles

CONTACTS AND LOCATIONS:
Overall Officials: Rowlens M. Melduni, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials